CLINICAL TRIAL: NCT05778981
Title: Endothelial Dysfunction During Non-cardiac Surgery and Major Clinical Events
Brief Title: Endothelial Dysfunction and Non-cardiac Surgery
Status: Recruiting | Type: Observational
Sponsor: University of Chile (Other)
Collaborators: Agencia Nacional de Investigación y Desarrollo (Other)
Responsible Party: Principal Investigator, Felipe Andrés Maldonado Caniulao, Principal Investigator, University of Chile
Other Study IDs: OAIC 1316/22
Record Dates: First submitted 2023-02-21; First posted 2023-03-22 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Surgery; Cardiac Death; Stroke; Myocardial Injury
Keywords: FMD; Flow-Mediated Dilatation; Troponin
MeSH Terms: conditions — Death; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: FMD - Troponin measurement — Echographic FMD evaluation. Pre and post-operative troponin measurements.

SUMMARY:
Endothelial dysfunction is a cardiovascular disease hallmark. After non-cardiac surgery, cardiovascular events correlate with surgical outcomes. Understanding the role of endothelial function in these events is crucial.

This research aims to study endothelial function and its association with cardiovascular events.

DETAILED DESCRIPTION:
To study the presence of endothelial damage and its association with cardiac events, the investigators will perform an observational study to evaluate flow-induced dilatation of the brachial artery in patients scheduled for non-cardiac surgery.

After ethical review board approval, the investigators will select 200 patients admitted for non-cardiac surgery. After the patient written consent, the investigators will perform an ultrasound evaluation of the brachial artery flow-mediated dilatation. This will be performed before, during, and after surgery. A basal troponin level will be obtained and repeatedly measured in the three days after surgery.

The investigators will observe clinical outcomes one, 3, and 6 months after the hospitalization.

To observe 8% of events, for a 5% alpha and 80% power, 161 patients are needed for our study. The authors considered that to account for a loss of 10% of patients, a sample of 177 patients will be required. Considering no national or local incidence of cardiovascular events, we aim to complete a 200-patient selection.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Patients 45 years or older

Exclusion Criteria:

* Refuse to participate in the study
* Myocardial injury or acute myocardial infarction less than two weeks ago
* Patients who expect less than 2 days of hospitalization
* Patients in whom the troponin elevation is attributed to a secondary cause (for example, sepsis, pulmonary thromboembolism, electrical cardioversion, etc.)
* Use of chemotherapy less than 2 weeks ago

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for non-cardiac surgery of 45 years old and older.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-03-25 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Major Cardiac Events | 7 days after surgery
  Result composed of myocardial infarction, cardiac arrest, and Death
Major Cardiac Events | 1 month after surgery
  Result composed of myocardial infarction, cardiac arrest, and Death
Major Cardiac Events | 3 months after surgery
  Result composed of myocardial infarction, cardiac arrest, and Death
Major Cardiac Events | 6 months after surgery
  Result composed of myocardial infarction, cardiac arrest, and Death

SECONDARY OUTCOMES:
Myocardial Injury | 1 day after surgery
  Troponin I elevation
Myocardial Injury | 2 days after surgery
  Troponin I elevation
Myocardial Injury | 3 days after surgery
  Troponin I elevation
Stroke | 7 days after surgery
  Stroke incidence after surgery
Stroke | 1 month after surgery
  Stroke incidence after surgery
Stroke | 3 months after surgery
  Stroke incidence after surgery
Stroke | 6 months after surgery
  Stroke incidence after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Maldonado||, M.D.,M.Sc., Study Chair — Hospital Clinico de la Universidad de Chile
Locations (1):
- Hospital Clínico de la Universidad de Chile, Independencia, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No